CLINICAL TRIAL: NCT01885260
Title: A Double Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of ISIS 449884 Administered Once Weekly to Patients With Type 2 Diabetes Mellitus Being Treated With Metformin
Brief Title: Safety, Tolerability and Efficacy of ISIS-GCGRRx in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 449884-CS2
Record Dates: First submitted 2013-06-13; First posted 2013-06-24 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ISIS-GCGRRx Dose Level 1 (Experimental): ISIS-GCGRRx Dose Level 1
  Interventions: Drug: ISIS-GCGRRx - Dose Level 1
- ISIS-GCGRRx Dose Level 2 (Experimental): ISIS-GCGRRx Dose Level 2
  Interventions: Drug: ISIS-GCGRRx - Dose Level 2
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS-GCGRRx - Dose Level 1 — 3 doses on alternate days during the first week and then once weekly for 12 weeks
  Other Names: Isis 449884
  Arms: ISIS-GCGRRx Dose Level 1
Drug: ISIS-GCGRRx - Dose Level 2 — 3 doses on alternate days during the first week and then once weekly for 12 weeks
  Other Names: Isis 449884
  Arms: ISIS-GCGRRx Dose Level 2
Drug: Placebo — 3 doses on alternate days during the first week and then once weekly for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of ISIS-GCGRRx in combination with metformin versus placebo + metformin

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 75
* BMI greater than or equal to 25
* HbA1c greater than or equal to 7.5% and less than or equal to 10.5%
* Type 2 Diabetes Mellitus and on stable dose of oral metformin
* Agree to conduct home-based (fasted) blood glucose testing as directed

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam
* Show evidence of uncorrected hypothyroidism or hyperthyroidism hormone results
* History of renal transplantation or renal dialysis
* History of liver disease
* History of greater than 3 episodes of severe hypoglycemia within 6 months of screening
* Use of oral anti-diabetic medication other than metformin within 3 months of screening
* History of diabetic ketoacidosis
* Any other significant illness or condition that may interfere with the patient participating or completing the study
* Inability or unwillingness to comply with protocol or study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The effect of ISIS-GCGRRx on serum fructosamine | 14 Weeks
  Change from Baseline to Week 14

SECONDARY OUTCOMES:
The safety of ISIS-GCGRRx | 25 Weeks
  By determining the incidence, severity, dose-relationship adverse effects, and changes in laboratory evaluations
The tolerability of ISIS-GCGRRx | 25 Weeks
  By determining the incidence, severity, dose-relationship adverse effects, and changes in laboratory evaluations

CONTACTS AND LOCATIONS:
Locations (24):
- United States (18):
  - Isis Investigational Site, Birmingham, Alabama
  - Isis Investigational Site, Muscle Shoals, Alabama
  - Isis Investigational Site, Anaheim, California
  - Isis Investigational Site, Chino, California
  - Isis Investigational Site, Los Angeles, California
  - Isis Investigational Site, DeLand, Florida
  - Isis Investigational Site, Fort Lauderdale, Florida
  - Isis Investigational Site, Miami, Florida
  - Isis Investigational Site, Marietta, Georgia
  - Isis Investigational Site, Las Vegas, Nevada
  - Isis Investigational Site, Cincinnati, Ohio
  - Isis Investigational Site, Oklahoma City, Oklahoma
  - Isis Investigational Site, Eugene, Oregon
  - Isis Investigational Site, Corpus Christi, Texas
  - Isis Investigational Site, Katy, Texas
  - Isis Investigational Site, Salt Lake City, Utah
  - Isis Investigational Site, Renton, Washington
  - Isis Investigational Site, Spokane, Washington
- South Africa (6):
  - Isis Investigational Site, Lenasia South, Gauteng
  - Isis Investigational Site, Soweto, Gauteng
  - Isis Investigational Site, Durban, KwaZulu-Natal
  - Isis Investigational Site, Cape Town, Western Cape
  - Isis Investigational Site, Parow, Cape Town, Western Cape
  - Isis Investigational Site, Western Cape, Western Cape

REFERENCES:
- [Derived] Morgan ES, Tai LJ, Pham NC, Overman JK, Watts LM, Smith A, Jung SW, Gajdosik M, Krssak M, Krebs M, Geary RS, Baker BF, Bhanot S. Antisense Inhibition of Glucagon Receptor by IONIS-GCGRRx Improves Type 2 Diabetes Without Increase in Hepatic Glycogen Content in Patients With Type 2 Diabetes on Stable Metformin Therapy. Diabetes Care. 2019 Apr;42(4):585-593. doi: 10.2337/dc18-1343. Epub 2019 Feb 14. PMID 30765435